CLINICAL TRIAL: NCT04989257
Title: 24-month Ticagrelor-based Dual-antiplatelet Therapy Versus Clopidogrel-based Dual-antiplatelet theRapy aftEr 12 Months of DrUg-eluting Stent Implantation in High isChEmic Risk Patients: P-REDUCE Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0591
Record Dates: First submitted 2021-07-01; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: High Ischemic Risk

STUDY DESIGN:
Intervention Model Description: Ticagrelor-based dual-antiplatelet therapy vs. Clopidogrel-based dual-antiplatelet therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor-based dual-antiplatelet therapy (Experimental): Aspirin with ticagrelor
  Interventions: Drug: Ticagrelor-based dual-antiplatelet therapy
- Clopidogrel-based dual-antiplatelet therapy (Active Comparator): Aspirin with clopidogrel
  Interventions: Drug: Clopidogrel-based dual-antiplatelet therapy

INTERVENTIONS:
Drug: Ticagrelor-based dual-antiplatelet therapy — Aspirin with ticagrelor
  Arms: Ticagrelor-based dual-antiplatelet therapy
Drug: Clopidogrel-based dual-antiplatelet therapy — Aspirin with clopidogrel
  Arms: Clopidogrel-based dual-antiplatelet therapy

SUMMARY:
The purpose of this prospective randomized clinical trial is to compare the clinical outcomes between aspirin with ticagrelor versus aspirin with clopidogrel in high ischemic risk patients beyond 12 months after percutaneous coronary intervention with drug-eluting stent implantation

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years old
2. History of drug-eluting stent implantation due to acute myocardial infarction 12 to 24 months ago
3. High-risk for ischemic events (at least one of the following) 1) Age >65 years old 2) Medical treatments for diabetes mellitus 3) Multi-vessel coronary artery disease 4) More than 2 episodes of myocardial infarction 5) Chronic kidney disease (stage III or IV)

Exclusion Criteria:

1. Age ≥85 years old
2. Pregnant women or women with potential childbearing
3. Life expectancy < 1 year
4. Inability to understand or read the informed consent
5. Need for long-term anticoagulation therapy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3488 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause death, myocardial infarction, or stroke | up to 24 months
  Composite of all-cause death, myocardial infarction, or stroke at 24 months after randomization

SECONDARY OUTCOMES:
BARC type 2, 3, or 5 bleeding | up to 24 months
  BARC type 2, 3, or 5 bleeding at 24 months after randomization
All-cause death | up to 24 months
  All-cause death at 24 months after randomization
Myocardial infarction | up to 24 months
  Myocardial infarction at 24 months after randomization
Stroke | up to 24 months
  Stroke at 24 months after randomization
Cardiac death | up to 24 months
  Cardiac death at 24 months after randomization
Composite of all-cause death, myocardial infarction, stroke, or BARC type 2, 3, or 5 bleeding | up to 24 months
  Composite of all-cause death, myocardial infarction, stroke, or BARC type 2, 3, or 5 bleeding at 24 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Byeong-Keuk Kim, Principal Investigator — Yonsei University
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No